CLINICAL TRIAL: NCT02996110
Title: A Phase 2, Real-time Assessment of Combination Therapies in Immuno-Oncology Study in Participants With Advanced Renal Cell Carcinoma (FRACTION-RCC)
Brief Title: A Study to Test Combination Treatments in People With Advanced Renal Cell Carcinoma
Acronym: FRACTION-RCC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA018-005; 2016-003082-26 (EudraCT Number)
Record Dates: First submitted 2016-12-15; First posted 2016-12-19 (Estimated); Results first posted 2022-12-19 (Actual); Last update posted 2022-12-19 (Actual); Status verified 2022-11

CONDITIONS: Advanced Cancer
MeSH Terms: interventions — Nivolumab; Ipilimumab; relatlimab; linrodostat; BMS-813160

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Nivolumab + Ipilimumab (Active Comparator): Nivolumab + Ipilimumab
  Interventions: Biological: Nivolumab; Biological: Ipilimumab
- Nivolumab + Relatlimab (Experimental): Nivolumab + Relatlimab
  Interventions: Biological: Nivolumab; Biological: Relatlimab
- Nivolumab + BMS-986205 (Experimental): Nivolumab + BMS-986205
  Interventions: Biological: Nivolumab; Drug: BMS-986205
- Nivolumab + BMS-813160 (Experimental): Nivolumab + BMS-813160 (CCR2/5 dual antagonist)
  Interventions: Biological: Nivolumab; Drug: BMS-813160

INTERVENTIONS:
Biological: Nivolumab — Specified Dose on Specified Days
  Other Names: Opdivo; BMS-936558
Biological: Ipilimumab — Specified Dose on Specified Days
  Other Names: BMS-734016; Yervoy
  Arms: Nivolumab + Ipilimumab
Biological: Relatlimab — Specified Dose on Specified Days
  Other Names: BMS-986016
  Arms: Nivolumab + Relatlimab
Drug: BMS-986205 — Specified Dose on Specified Days
  Arms: Nivolumab + BMS-986205
Drug: BMS-813160 — Specified Dose on Specified Days
  Arms: Nivolumab + BMS-813160

SUMMARY:
The purpose of this study is to test the effectiveness and safety of various nivolumab combinations compared to nivolumab and ipilimumab in participants with advanced kidney cancer

ELIGIBILITY:
Inclusion Criteria:

* Advanced Renal Cell Carcinoma
* Must have at least 1 lesion with measurable disease
* Life expectancy of at least 3 months
* Karnofsky Performance Status (KPS) must be =>70%

Exclusion Criteria:

* Patients/subjects with suspected or known central nervous system metastases unless adequately treated
* Patients/subjects with autoimmune disease
* Patients/subjects who need daily oxygen therapy

Other protocol defined inclusion/exclusion criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 182 (Actual)
Dates: Start 2017-02-02 (Actual); Primary Completion 2021-11-23 (Actual); Study Completion 2021-11-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (32):
- United States (20):
  - Local Institution - 0037, New Haven, Connecticut
  - Local Institution, Tampa, Florida
  - Local Institution - 0031, Augusta, Georgia
  - Local Institution - 0006, Chicago, Illinois
  - Local Institution - 0007, Baltimore, Maryland
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - Local Institution - 0011, Detroit, Michigan
  - Local Institution - 0008, St Louis, Missouri
  - Roswell Park Cancer Institute, Buffalo, New York
  - Local Institution - 0005, New York, New York
  - Local Institution - 0043, Charlotte, North Carolina
  - Local Institution - 0014, Columbus, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - Local Institution - 0002, Allentown, Pennsylvania
  - Hollings Cancer Center, Charleston, South Carolina
  - Local Institution - 0025, Nashville, Tennessee
  - Ut Southwestern Medical Center, Dallas, Texas
  - Local Institution - 0024, Charlottesville, Virginia
  - University of Washington - Seattle Cancer Care Alliance, Seattle, Washington
- Australia (2):
  - Local Institution - 0032, Westmead, New South Wales
  - Monash Medical Centre Clayton, Bentleigh, Victoria
- Local Institution - 0044, Linz, Upper Austria, Austria
- Canada (5):
  - Local Institution - 0038, Hamilton, Ontario
  - Local Institution - 0029, Oshawa, Ontario
  - Local Institution - 0035, Toronto, Ontario
  - Local Institution - 0034, Montreal, Quebec
  - Local Institution - 0030, Québec, Quebec
- Israel (2):
  - Local Institution, Haifa
  - Local Institution, Ramat Gan
- Italy (2):
  - Local Institution - 0010, Milan
  - Local Institution - 0012, Napoli

REFERENCES:
- [Derived] Choueiri TK, Kluger H, George S, Tykodi SS, Kuzel TM, Perets R, Nair S, Procopio G, Carducci MA, Castonguay V, Folefac E, Lee CH, Hotte SJ, Miller WH Jr, Saggi SS, Lee CW, Desilva H, Bhagavatheeswaran P, Motzer RJ, Escudier B. FRACTION-RCC: nivolumab plus ipilimumab for advanced renal cell carcinoma after progression on immuno-oncology therapy. J Immunother Cancer. 2022 Nov;10(11):e005780. doi: 10.1136/jitc-2022-005780. PMID 36328377
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.BMSStudyConnect.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of the 178 participants that were treated, 60 were initially randomized to Track 1 and 118 were initially randomized to Track 2. The 152 participants that started treatment in Track 2 include the total number of participants that received treatment in each arm which incorporates the 35 participants from Track 1 or 2 that were re-randomized to receive a different treatment combination in Track 2.
Groups:
- Arm 1: Nivolumab Plus Ipilimumab (BMS-734016): Nivolumab was administered at 3 mg/kg via IV infusion followed by ipilimumab 1 mg/kg administered IV over approximately 30 minutes every 3 weeks for 4 doses. Six weeks after the last dose of combination study treatment nivolumab 480 mg was administered IV over approximately 30 minutes every 4 weeks until completion of approximately 2 years of study treatment, clinical deterioration suggesting that no further benefit from study treatment is likely, intolerable toxicity, meeting of criteria for discontinuation of study treatment, or withdrawal of consent, whichever occurred first.
- Arm 2: Nivolumab Plus Relatlimab (BMS-986016): Nivolumab was administered at a flat dose of 240 mg via IV infusion every 2 weeks followed by 80 mg BMS-986016 administered IV approximately 60 minutes every 2 weeks until completion of approximately 2 years of study treatment, clinical deterioration suggesting that no further benefit from study treatment is likely, intolerable toxicity, meeting of criteria for discontinuation of study treatment, or withdrawal of consent, whichever occurred first.
- Arm 3: Nivolumab Plus BMS-986205: Nivolumab was administered as a flat dose of 480 mg via IV infusion every 4 weeks, and BMS-986205 taken orally at a dose of 100 mg daily for up to 2 years, clinical deterioration suggesting that no further benefit from study treatment is likely, intolerable toxicity, meeting of criteria for discontinuation of study treatment, or withdrawal of consent, whichever occurred first.
- Arm 4: Nivolumab Plus BMS-813160 150 mg: Nivolumab was administered as a flat dose of 480 mg by IV infusion every 4 weeks combined with oral BMS-813160, 150 mg daily for up to 2 years, clinical deterioration suggesting that no further benefit from study treatment is likely, intolerable toxicity, meeting of criteria for discontinuation of study treatment, or withdrawal of consent, whichever occurred first.
- Arm 5: Nivolumab Plus BMS-813160 300mg: Nivolumab was administered as a flat dose of 480 mg by IV infusion every 4 weeks combined with oral BMS-813160, 300 mg twice daily for up to 2 years, clinical deterioration suggesting that no further benefit from study treatment is likely, intolerable toxicity, meeting of criteria for discontinuation of study treatment, or withdrawal of consent, whichever occurred first.
Period: Pre-Treatment
Arm/Group | Arm 1: Nivolumab Plus Ipilimumab (BMS-734016) | Arm 2: Nivolumab Plus Relatlimab (BMS-986016) | Arm 3: Nivolumab Plus BMS-986205 | Arm 4: Nivolumab Plus BMS-813160 150 mg | Arm 5: Nivolumab Plus BMS-813160 300mg
Started (Initial Randomization) | 65 | 56 | 26 | 17 | 18
Completed (Continuing Into Treatment Period) | 65 | 55 | 25 | 17 | 16
Not Completed | 0 | 1 | 1 | 0 | 2
Not completed — Other Reasons | 0 | 1 | 0 | 0 | 1
Not completed — Participant Withdrew Consent | 0 | 0 | 1 | 0 | 1
Period: Track 1
Arm/Group | Arm 1: Nivolumab Plus Ipilimumab (BMS-734016) | Arm 2: Nivolumab Plus Relatlimab (BMS-986016) | Arm 3: Nivolumab Plus BMS-986205 | Arm 4: Nivolumab Plus BMS-813160 150 mg | Arm 5: Nivolumab Plus BMS-813160 300mg
Started | 30 | 30 | 0 | 0 | 0
Re-Randomized to Track 2 | 5 | 6 | 0 | 0 | 0
Completed | 7 | 8 | 0 | 0 | 0
Not Completed | 23 | 22 | 0 | 0 | 0
Not completed — Disease Progression | 15 | 17 | 0 | 0 | 0
Not completed — Adverse Event Unrelated to Study Drug | 1 | 1 | 0 | 0 | 0
Not completed — Study Drug Toxicity | 5 | 3 | 0 | 0 | 0
Not completed — Participant Requested to Discontinue Study Treatment | 1 | 0 | 0 | 0 | 0
Not completed — Administrative Reason by Sponsor | 0 | 1 | 0 | 0 | 0
Not completed — Participant no Longer Met Study Criteria | 1 | 0 | 0 | 0 | 0
Period: Track 2
Arm/Group | Arm 1: Nivolumab Plus Ipilimumab (BMS-734016) | Arm 2: Nivolumab Plus Relatlimab (BMS-986016) | Arm 3: Nivolumab Plus BMS-986205 | Arm 4: Nivolumab Plus BMS-813160 150 mg | Arm 5: Nivolumab Plus BMS-813160 300mg
Started | 46 | 32 | 31 | 21 | 22
No Pre-Randomization | 35 | 25 | 25 | 17 | 16
Re-Randomized From Track 1 Nivolumab + Relatlimab | 2 | 0 | 2 | 1 | 1
Re-Randomized From Track 1 Nivolumab + Ipilimumab | 0 | 3 | 1 | 1 | 0
Re-Randomized From Track 2 Nivolumab + Relatlimab | 7 | 0 | 2 | 0 | 1
Re-Randomized From Track 2 Nivolumab + BMS986205 | 2 | 2 | 0 | 1 | 2
Previously Un-Treated But Re-Randomized | 0 | 0 | 0 | 1 | 0
Re-Randomized From Track 2 Nivolumab + Ipilimumab | 0 | 2 | 1 | 0 | 2
Completed | 4 | 3 | 1 | 1 | 1
Not Completed | 42 | 29 | 30 | 20 | 21
Not completed — Disease Progression | 33 | 26 | 19 | 16 | 15
Not completed — Adverse Event Unrelated to Study Drug | 4 | 0 | 0 | 1 | 1
Not completed — Death | 0 | 0 | 1 | 0 | 1
Not completed — Study Drug Toxicity | 4 | 1 | 4 | 1 | 0
Not completed — Participant Requested to Discontinue Study Treatment | 0 | 0 | 2 | 1 | 2
Not completed — Participant Withdrew Consent | 1 | 2 | 3 | 1 | 1
Not completed — Other Reasons | 0 | 0 | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Arms 1 and 2 take into account both Track 1 and Track 2 participants as well as those rerandomized to the respective arms in Track 2.
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1: Nivolumab Plus Ipilimumab (BMS-734016) | Arm 2: Nivolumab Plus Relatlimab (BMS-986016) | Arm 3: Nivolumab Plus BMS-986205 | Arm 4: Nivolumab Plus BMS-813160 150 mg | Arm 5: Nivolumab Plus BMS-813160 300mg | Total
Number analyzed (Participants) | 65 | 56 | 26 | 17 | 18 | 182
Age, Categorical [Count of Participants; unit: Participants] — Population: The analysis population consists of all participants treated (including those re-randomized) in each Arm.
  Participants
    <=18 years | 0 | 0 | 0 | 0 | 0 | 0
    Between 18 and 65 years | 40 | 41 | 16 | 12 | 11 | 120
    >=65 years | 25 | 15 | 10 | 5 | 7 | 62
Sex: Female, Male [Count of Participants; unit: Participants] — Population: The analysis population consists of all participants treated (including those re-randomized) in each Arm.
  Participants
    Female | 14 | 16 | 6 | 4 | 9 | 49
    Male | 51 | 40 | 20 | 13 | 9 | 133
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: The analysis population consists of all participants treated (including those re-randomized) in each Arm.
  Participants
    Track 2: Hispanic or Latino | 3 | 2 | 2 | 1 | 0 | 8
    Track 2: Not Hispanic or Latino | 37 | 34 | 19 | 12 | 10 | 112
    Track 2: Unknown or Not Reported | 25 | 20 | 5 | 4 | 8 | 62
Race/Ethnicity, Customized [Number; unit: Participants] — Population: The analysis population consists of all participants treated (including those re-randomized) in each Arm.
  Participants
    White | 62 | 52 | 23 | 14 | 17 | 168
    Asian Indian | 1 | 0 | 0 | 0 | 0 | 1
    Chinese | 0 | 1 | 0 | 0 | 0 | 1
    Asian Other | 1 | 1 | 0 | 0 | 0 | 2
    Other | 1 | 2 | 2 | 2 | 0 | 7
    Black or African American | 0 | 0 | 1 | 1 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR) Per Investigator
Description: ORR is percent of participants whose best overall response (BOR) is complete response (CR) or partial response (PR).
  BOR is the best response from the start of the study treatment until objectively documented progression per RECIST v1.1 or subsequent anticancer therapy, whichever occurs first.
  For participants who received re-treatment or were re-randomized, the re-treatment and re-randomized therapies were considered subsequent anticancer therapy.
  CR is the disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) have reduction in short axis to <10 mm.
  PR is at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
  The Response Evaluation Criteria in Solid Tumors (RECIST) is a standard way to measure the response of a tumor to treatment.
  CR+PR, confidence interval based on Clopper and Pearson method.
Time Frame: From first dose of study treatment until progression or subsequent anticancer therapy, whichever occurs first (assessed up to approximately 247 weeks)
Population: All treated participants. Some participants were re-randomized to receive multiple treatment options during the course of the study.
Measure: Number (95% Confidence Interval); unit: Percent of participants
Arm/Group | Arm 1: Nivolumab Plus Ipilimumab (BMS-734016) | Arm 2: Nivolumab Plus Relatlimab (BMS-986016) | Arm 3: Nivolumab Plus BMS-986205 | Arm 4: Nivolumab Plus BMS-813160 150 mg | Arm 5: Nivolumab Plus BMS-813160 300mg
Number analyzed (Participants) | 76 | 62 | 31 | 21 | 22
Percent of participants
  Track 1: number analyzed (Participants) | 30 | 30 | 0 | 0 | 0
  Track 1 | 20 [7.7 to 38.6] | 30 [14.7 to 49.4] |  |  |
  Track 2: number analyzed (Participants) | 46 | 32 | 31 | 21 | 22
  Track 2 | 17.4 [7.8 to 31.4] | 3.1 [0.1 to 16.2] | 3.2 [0.1 to 16.7] | 9.5 [1.2 to 30.4] | 0.0 [0.0 to 15.4]

2. Primary Outcome: Median Duration of Response (DOR) Per Investigator
Description: Duration of Response is defined as the time between the date of first response and the date of first documented disease progression as determined by RECIST 1.1 or death due to any cause (death occurring after re-treatment or randomization to new combination treatment was not considered), whichever occurred first.
  Complete Response (CR) is the disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm.
  Partial Response (PR) is at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
  Median computed using Kaplan -Meier method
Time Frame: From first dose to the date of first documented disease progression or death due to any cause (assessed from an average of 22 weeks up to approximately 247 weeks)
Population: All treated participants with a best overall response of CR or PR. Some participants were re-randomized to receive multiple treatment options during the course of the study.
Measure: Median (Full Range); unit: Weeks
Arm/Group | Arm 1: Nivolumab Plus Ipilimumab (BMS-734016) | Arm 2: Nivolumab Plus Relatlimab (BMS-986016) | Arm 3: Nivolumab Plus BMS-986205 | Arm 4: Nivolumab Plus BMS-813160 150 mg | Arm 5: Nivolumab Plus BMS-813160 300mg
Number analyzed (Participants) | 14 | 10 | 1 | 2 | 0
Weeks
  Track 1: number analyzed (Participants) | 6 | 9 | 0 | 0 | 0
  Track 1 | NA [33.4 to 139.9] — Insufficient number of participants with events. Five of the 6 participants received subsequent therapy prior to progression or death, thus their DOR was censored at the last tumor assessment. | 32.57 [0.1 to 52.6] |  |  |
  Track 2: number analyzed (Participants) | 8 | 1 | 1 | 2 | 0
  Track 2 | 68.00 [0.1 to 117.6] | 99.4 [99.4 to 99.4] | NA [NA to NA] — Insufficient number of participants with events | NA [NA to NA] — Insufficient number of participants with events |

3. Primary Outcome: Progression Free Survival Rate (PFSR) at 24 Weeks.
Description: The PFSR at 24 weeks is defined as the proportion of treated participants remaining progression free and surviving at 24 weeks since the first dosing date.
  Progressive Disease (PD) is at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. (Note: the appearance of one or more new lesions is also considered progression).
  Point estimates are derived from Kaplan-Meier analyses, the 95% CIs are derived from Greenwood formula
Time Frame: 24 weeks after first treatment dose.
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Proportion of participants
Arm/Group | Arm 1: Nivolumab Plus Ipilimumab (BMS-734016) | Arm 2: Nivolumab Plus Relatlimab (BMS-986016) | Arm 3: Nivolumab Plus BMS-986205 | Arm 4: Nivolumab Plus BMS-813160 150 mg | Arm 5: Nivolumab Plus BMS-813160 300mg
Number analyzed (Participants) | 76 | 62 | 31 | 21 | 22
Proportion of participants
  Track 1: number analyzed (Participants) | 30 | 30 | 0 | 0 | 0
  Track 1 | 0.491 [0.294 to 0.661] | 0.429 [0.246 to 0.600] |  |  |
  Track 2: number analyzed (Participants) | 46 | 32 | 31 | 21 | 22
  Track 2 | 0.432 [0.277 to 0.577] | 0.194 [0.079 to 0.346] | 0.278 [0.118 to 0.464] | 0.468 [0.237 to 0.670] | NA [NA to NA] — Insufficient number of participants with events.

4. Secondary Outcome: Number of Participants With Adverse Events (AEs)
Description: An Adverse Event (AE) is defined as any new untoward medical occurrence or worsening of a preexisting medical condition in a clinical investigation participant administered study treatment and that does not necessarily have a causal relationship with this treatment.
Time Frame: From first dose to 100 days after last dose of study therapy (assessed up to approximately 118 weeks)
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Arm 1: Nivolumab Plus Ipilimumab (BMS-734016) | Arm 2: Nivolumab Plus Relatlimab (BMS-986016) | Arm 3: Nivolumab Plus BMS-986205 | Arm 4: Nivolumab Plus BMS-813160 150 mg | Arm 5: Nivolumab Plus BMS-813160 300mg
Number analyzed (Participants) | 76 | 62 | 31 | 21 | 22
Participants
  Track 1: number analyzed (Participants) | 30 | 30 | 0 | 0 | 0
  Track 1 | 29 | 30 |  |  |
  Track 2: number analyzed (Participants) | 46 | 32 | 31 | 21 | 22
  Track 2 | 45 | 32 | 31 | 19 | 21

5. Secondary Outcome: Number of Participants With Serious Adverse Events (SAEs)
Description: Serious Adverse Event (SAE) is defined as any untoward medical occurrence that, at any dose results in death, is life-threatening (defined as an event in which the participant was at risk of death at the time of the event; it does not refer to an event which hypothetically might have caused death if it were more severe), requires inpatient hospitalization or causes prolongation of existing hospitalization
Time Frame: From first dose to 100 days after last dose of study therapy (assessed up to approximately 118 weeks)
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Arm 1: Nivolumab Plus Ipilimumab (BMS-734016) | Arm 2: Nivolumab Plus Relatlimab (BMS-986016) | Arm 3: Nivolumab Plus BMS-986205 | Arm 4: Nivolumab Plus BMS-813160 150 mg | Arm 5: Nivolumab Plus BMS-813160 300mg
Number analyzed (Participants) | 76 | 62 | 31 | 21 | 22
Participants
  Track 1: number analyzed (Participants) | 30 | 30 | 0 | 0 | 0
  Track 1 | 17 | 15 |  |  |
  Track 2: number analyzed (Participants) | 46 | 32 | 31 | 21 | 22
  Track 2 | 28 | 16 | 16 | 9 | 15

6. Secondary Outcome: Number of Participants With Adverse Events (AEs) Leading to Discontinuation
Description: as for outcome 4
Time Frame: From first dose to 100 days after last dose of study therapy (assessed up to approximately 118 weeks)
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Arm 1: Nivolumab Plus Ipilimumab (BMS-734016) | Arm 2: Nivolumab Plus Relatlimab (BMS-986016) | Arm 3: Nivolumab Plus BMS-986205 | Arm 4: Nivolumab Plus BMS-813160 150 mg | Arm 5: Nivolumab Plus BMS-813160 300mg
Number analyzed (Participants) | 76 | 62 | 31 | 21 | 22
Participants
  Track 1: number analyzed (Participants) | 30 | 30 | 0 | 0 | 0
  Track 1 | 7 | 7 |  |  |
  Track 2: number analyzed (Participants) | 46 | 32 | 31 | 21 | 22
  Track 2 | 10 | 3 | 6 | 2 | 4

7. Secondary Outcome: Number of Participants Who Died
Description: Death is defined as the cessation of all vital functions of the body including the heartbeat, brain activity (including the brain stem), and breathing.
Time Frame: From first dose to 100 days after last dose of study therapy (assessed up to approximately 118 weeks)
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Arm 1: Nivolumab Plus Ipilimumab (BMS-734016) | Arm 2: Nivolumab Plus Relatlimab (BMS-986016) | Arm 3: Nivolumab Plus BMS-986205 | Arm 4: Nivolumab Plus BMS-813160 150 mg | Arm 5: Nivolumab Plus BMS-813160 300mg
Number analyzed (Participants) | 76 | 62 | 31 | 21 | 22
Participants
  Track 1: number analyzed (Participants) | 30 | 30 | 0 | 0 | 0
  Track 1 | 12 | 15 |  |  |
  Track 2: number analyzed (Participants) | 46 | 32 | 31 | 21 | 22
  Track 2 | 27 | 17 | 13 | 10 | 13

8. Secondary Outcome: Number of Participants With Abnormal Thyroid Test Results - Track 1
Description: The number of participants with laboratory abnormalities in specific thyroid tests based on SI conventional units. TSH = Thyroid Stimulating Hormone LLN = Lower Limit of Normal ULN = Upper Limit of Normal.
Time Frame: From first dose to 30 days after last dose of study therapy (approximately 108 weeks)
Population: All treated participants with at least one on-treatment TSH measurement
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1: Nivolumab Plus Ipilimumab (BMS-734016) | Arm 2: Nivolumab Plus Relatlimab (BMS-986016) | Arm 3: Nivolumab Plus BMS-986205 | Arm 4: Nivolumab Plus BMS-813160 150 mg | Arm 5: Nivolumab Plus BMS-813160 300mg
Number analyzed (Participants) | 28 | 27 | 0 | 0 | 0
Participants
  TSH > ULN | 8 | 8 | 0 | 0 | 0
  TSH > ULN WITH TSH <= ULN AT BASELINE | 5 | 8 | 0 | 0 | 0
  TSH >ULN WITH ATLEAST ONE FT3/FT4 TEST VALUE <LLN | 3 | 3 | 0 | 0 | 0
  TSH >ULN WITH ALL OTHER FT3/FT4 TEST VALUES >= LLN | 3 | 2 | 0 | 0 | 0
  TSH > ULN WITH FT3/FT4 TEST MISSING | 2 | 3 | 0 | 0 | 0
  TSH < LLN | 10 | 5 | 0 | 0 | 0
  TSH <LLN WITH TSH >= LLN AT BASELINE | 9 | 5 | 0 | 0 | 0
  TSH <LLN WITH ATLEAST ONE FT3/FT4 TEST VALUE > ULN | 3 | 0 | 0 | 0 | 0
  TSH <LLN WITH ALL OTHER FT3/FT4 TEST VALUES <= ULN | 2 | 1 | 0 | 0 | 0
  TSH < LLN WITH FT3/FT4 TEST MISSING | 5 | 4 | 0 | 0 | 0

9. Secondary Outcome: Number of Participants With Abnormal Thyroid Test Results - Track 2
Description: as for outcome 8
Time Frame: From first dose to 30 days after last dose of study therapy (approximately 108 weeks)
Population: All treated participants with at Least One On-Treatment TSH measurement. Some participants were re-randomized to receive multiple treatment options during the course of the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1: Nivolumab Plus Ipilimumab (BMS-734016) | Arm 2: Nivolumab Plus Relatlimab (BMS-986016) | Arm 3: Nivolumab Plus BMS-986205 | Arm 4: Nivolumab Plus BMS-813160 150 mg | Arm 5: Nivolumab Plus BMS-813160 300mg
Number analyzed (Participants) | 42 | 30 | 25 | 17 | 13
Participants
  TSH > ULN | 14 | 14 | 6 | 3 | 4
  TSH > ULN WITH TSH <= ULN AT BASELINE | 8 | 6 | 3 | 2 | 2
  TSH >ULN WITH ATLEAST ONE FT3/FT4 TEST VALUE <LLN | 5 | 3 | 1 | 1 | 0
  TSH >ULN WITH ALL OTHER FT3/FT4 TEST VALUES >= LLN | 5 | 4 | 3 | 2 | 3
  TSH > ULN WITH FT3/FT4 TEST MISSING | 4 | 7 | 2 | 0 | 1
  TSH < LLN | 4 | 5 | 2 | 2 | 1
  TSH <LLN WITH TSH >= LLN AT BASELINE | 2 | 4 | 1 | 2 | 1
  TSH <LLN WITH ATLEAST ONE FT3/FT4 TEST VALUE > ULN | 1 | 0 | 1 | 1 | 0
  TSH <LLN WITH ALL OTHER FT3/FT4 TEST VALUES <= ULN | 0 | 3 | 0 | 0 | 0
  TSH < LLN WITH FT3/FT4 TEST MISSING | 3 | 2 | 1 | 1 | 1

10. Secondary Outcome: Number of Participants With Abnormal Hepatic Test Results - Track 1
Description: The number of participants with laboratory abnormalities in specific liver tests based on SI conventional units. ALT = Alanine Aminotransferase AST = Aspartate Aminotransferase ULN = Upper Limit of Normal
Time Frame: From first dose to 30 days after last dose of study therapy (approximately 108 weeks)
Population: All treated participants with at least one on-treatment AST, ALT and/or bilirubin test measurement
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1: Nivolumab Plus Ipilimumab (BMS-734016) | Arm 2: Nivolumab Plus Relatlimab (BMS-986016) | Arm 3: Nivolumab Plus BMS-986205 | Arm 4: Nivolumab Plus BMS-813160 150 mg | Arm 5: Nivolumab Plus BMS-813160 300mg
Number analyzed (Participants) | 28 | 30 | 0 | 0 | 0
Participants
  ALT OR AST > 3XULN | 2 | 4 | 0 | 0 | 0
  ALT OR AST> 5XULN | 1 | 2 | 0 | 0 | 0
  ALT OR AST> 10XULN | 0 | 0 | 00 | 0 | 0
  ALT OR AST > 20XULN | 0 | 0 | 0 | 0 | 0
  TOTAL BILIRUBIN > 2XULN | 0 | 0 | 0 | 0 | 0
  ALT/AST ELEV>3XULN;TOTAL BILIRUBIN>2XULN IN 1 DAY | 0 | 0 | 0 | 0 | 0
  ALT/AST ELEV>3XULN;TOTAL BILIRUBIN>2XULN IN 30 DAYS | 0 | 0 | 0 | 0 | 0

11. Secondary Outcome: Number of Participants With Abnormal Hepatic Test Results - Track 2
Description: as for outcome 10
Time Frame: From first dose to 30 days after last dose of study therapy (approximately 108 weeks)
Population: All treated participants with at least one on-treatment AST, ALT and/or bilirubin test measurement. Some participants were re-randomized to receive multiple treatment options during the course of the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1: Nivolumab Plus Ipilimumab (BMS-734016) | Arm 2: Nivolumab Plus Relatlimab (BMS-986016) | Arm 3: Nivolumab Plus BMS-986205 | Arm 4: Nivolumab Plus BMS-813160 150 mg | Arm 5: Nivolumab Plus BMS-813160 300mg
Number analyzed (Participants) | 44 | 32 | 29 | 17 | 18
Participants
  ALT OR AST > 3XULN | 3 | 1 | 1 | 0 | 0
  ALT OR AST> 5XULN | 2 | 0 | 1 | 0 | 0
  ALT OR AST> 10XULN | 0 | 0 | 0 | 0 | 0
  ALT OR AST > 20XULN | 0 | 0 | 0 | 0 | 0
  TOTAL BILIRUBIN > 2XULN | 2 | 0 | 0 | 0 | 0
  ALT/AST ELEV>3XULN;TOTAL BILIRUBIN>2XULN IN 1 DAY | 0 | 0 | 0 | 0 | 0
  ALT/AST ELEV>3XULN;TOTAL BILIRUBIN>2XULN IN 30 DAYS | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Participants were assessed for All-Cause Mortality from the date of their randomization until study completion (assessed up to approximately 250 weeks). SAEs and Other AEs were assessed from first dose to 100 days after last dose of study therapy (assessed up to approximately 118 weeks).
Description: The number at Risk for All-Cause Mortality represents all Randomized Participants. The number at Risk for Serious Adverse Events and Other (Not Including Serious) Adverse Events represents all participants that received at least 1 dose of study medication.
Groups:
- Track 1: Nivolumab Plus Ipilimumab (BMS-734016); Track 2: Nivolumab Plus Ipilimumab (BMS-734016): Nivolumab was administered at 3 mg/kg via IV infusion followed by ipilimumab 1 mg/kg administered IV over approximately 30 minutes every 3 weeks for 4 doses. Six weeks after the last dose of combination study treatment nivolumab 480 mg was administered IV over approximately 30 minutes every 4 weeks until completion of approximately 2 years of study treatment, clinical deterioration suggesting that no further benefit from study treatment is likely, intolerable toxicity, meeting of criteria for discontinuation of study treatment, or withdrawal of consent, whichever occurred first.
- Track 1: Nivolumab Plus Relatlimab (BMS-986016); Track 2: Nivolumab Plus Relatlimab (BMS-986016): Nivolumab was administered at a flat dose of 240 mg via IV infusion every 2 weeks followed by 80 mg BMS-986016 administered IV approximately 60 minutes every 2 weeks until completion of approximately 2 years of study treatment, clinical deterioration suggesting that no further benefit from study treatment is likely, intolerable toxicity, meeting of criteria for discontinuation of study treatment, or withdrawal of consent, whichever occurred first.
- Track 2: Nivolumab Plus BMS-986205: Nivolumab was administered as a flat dose of 480 mg via IV infusion every 4 weeks, and BMS-986205 taken orally at a dose of 100 mg daily for up to 2 years, clinical deterioration suggesting that no further benefit from study treatment is likely, intolerable toxicity, meeting of criteria for discontinuation of study treatment, or withdrawal of consent, whichever occurred first.
- Track 2: Nivolumab Plus BMS-813160 150 mg: Nivolumab was administered as a flat dose of 480 mg by IV infusion every 4 weeks combined with oral BMS-813160, 150 mg daily for up to 2 years, clinical deterioration suggesting that no further benefit from study treatment is likely, intolerable toxicity, meeting of criteria for discontinuation of study treatment, or withdrawal of consent, whichever occurred first.
- Track 2: Nivolumab Plus BMS-813160 300 mg: Nivolumab was administered as a flat dose of 480 mg by IV infusion every 4 weeks combined with oral BMS-813160, 300 mg twice daily for up to 2 years, clinical deterioration suggesting that no further benefit from study treatment is likely, intolerable toxicity, meeting of criteria for discontinuation of study treatment, or withdrawal of consent, whichever occurred first.
Arm/Group | Track 1: Nivolumab Plus Ipilimumab (BMS-734016) | Track 1: Nivolumab Plus Relatlimab (BMS-986016) | Track 2: Nivolumab Plus Ipilimumab (BMS-734016) | Track 2: Nivolumab Plus Relatlimab (BMS-986016) | Track 2: Nivolumab Plus BMS-986205 | Track 2: Nivolumab Plus BMS-813160 150 mg | Track 2: Nivolumab Plus BMS-813160 300 mg
All-Cause Mortality (participants affected / at risk) | 12/30 | 15/31 | 27/46 | 17/32 | 13/32 | 10/21 | 13/24
Serious Adverse Events (participants affected / at risk) | 17/30 | 15/30 | 28/46 | 16/32 | 16/31 | 9/21 | 15/22
Other Adverse Events (participants affected / at risk) | 28/30 | 29/30 | 42/46 | 31/32 | 29/31 | 18/21 | 17/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Track 1: Nivolumab Plus Ipilimumab (BMS-734016) (N=30) | Track 1: Nivolumab Plus Relatlimab (BMS-986016) (N=30) | Track 2: Nivolumab Plus Ipilimumab (BMS-734016) (N=46) | Track 2: Nivolumab Plus Relatlimab (BMS-986016) (N=32) | Track 2: Nivolumab Plus BMS-986205 (N=31) | Track 2: Nivolumab Plus BMS-813160 150 mg (N=21) | Track 2: Nivolumab Plus BMS-813160 300 mg (N=22)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Angina pectoris (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 1 | 0 | 0 | 1 | 0 | 0
Cardiac arrest (Cardiac disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 1 | 0 | 1 | 0 | 0 | 1 | 0
Myocarditis (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pericarditis (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Ventricular tachycardia (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Adrenal insufficiency (Endocrine disorders) | 1 | 0 | 0 | 1 | 1 | 0 | 0
Immune-mediated adrenal insufficiency (Endocrine disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Colitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Enteritis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Enterocolitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Large intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Lip swelling (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Mouth haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0
Oesophagitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Small intestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 1 | 0 | 0
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Fatigue (General disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0
General physical health deterioration (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0
Pain (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1
Biliary obstruction (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0
Hepatotoxicity (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Device related infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Epididymitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 4 | 0 | 0 | 3 | 2 | 0 | 2
Pneumonia influenzal (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pulmonary sepsis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Sialoadenitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 1
Urosepsis (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Wound infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Acetabulum fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Post procedural haematuria (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Wound dehiscence (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 2 | 0 | 0
Amylase increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Blood potassium increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Lipase increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Transaminases increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Failure to thrive (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 2 | 3 | 2 | 0 | 1 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Autoimmune myositis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0 | 1 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 2 | 0 | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0
Polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 1 | 1
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 5 | 6 | 5 | 3 | 1 | 4
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 1 | 0 | 0
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Metastatic renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Aphasia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Brain oedema (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Encephalopathy (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Facial paralysis (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Immune-mediated neuropathy (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Neuralgia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pyramidal tract syndrome (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Seizure (Nervous system disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0
Spinal cord compression (Nervous system disorders) | 0 | 2 | 1 | 1 | 1 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 1
Bladder perforation (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Immune-mediated nephritis (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Oliguria (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Renal haematoma (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 2 | 2 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 2 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 2 | 0 | 0
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Intertrigo (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Embolism (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Haematoma (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypotension (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Lymphoedema (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Track 1: Nivolumab Plus Ipilimumab (BMS-734016) (N=30) | Track 1: Nivolumab Plus Relatlimab (BMS-986016) (N=30) | Track 2: Nivolumab Plus Ipilimumab (BMS-734016) (N=46) | Track 2: Nivolumab Plus Relatlimab (BMS-986016) (N=32) | Track 2: Nivolumab Plus BMS-986205 (N=31) | Track 2: Nivolumab Plus BMS-813160 150 mg (N=21) | Track 2: Nivolumab Plus BMS-813160 300 mg (N=22)
Anaemia (Blood and lymphatic system disorders) | 8 | 5 | 8 | 4 | 4 | 2 | 2
Sinus tachycardia (Cardiac disorders) | 1 | 1 | 0 | 1 | 2 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 2 | 1 | 1 | 0 | 1 | 0
Hyperthyroidism (Endocrine disorders) | 4 | 3 | 0 | 0 | 1 | 0 | 1
Hypothyroidism (Endocrine disorders) | 4 | 6 | 2 | 0 | 3 | 0 | 0
Dry eye (Eye disorders) | 1 | 0 | 0 | 3 | 0 | 0 | 0
Vision blurred (Eye disorders) | 2 | 2 | 0 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 3 | 1 | 5 | 4 | 2 | 1 | 1
Colitis (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 3 | 8 | 5 | 12 | 6 | 2 | 2
Diarrhoea (Gastrointestinal disorders) | 6 | 9 | 14 | 7 | 5 | 6 | 1
Dry mouth (Gastrointestinal disorders) | 1 | 4 | 4 | 1 | 0 | 0 | 1
Epigastric discomfort (Gastrointestinal disorders) | 1 | 0 | 0 | 2 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 3 | 1 | 2 | 1 | 0
Nausea (Gastrointestinal disorders) | 10 | 7 | 14 | 8 | 8 | 6 | 4
Oral pain (Gastrointestinal disorders) | 0 | 0 | 2 | 2 | 0 | 2 | 1
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 6 | 3 | 1 | 4 | 0
Vomiting (Gastrointestinal disorders) | 5 | 6 | 7 | 2 | 6 | 2 | 0
Asthenia (General disorders) | 2 | 0 | 3 | 2 | 3 | 2 | 1
Chest discomfort (General disorders) | 1 | 0 | 0 | 1 | 0 | 2 | 0
Chills (General disorders) | 3 | 2 | 4 | 3 | 0 | 0 | 0
Fatigue (General disorders) | 9 | 13 | 15 | 11 | 8 | 7 | 6
Gait disturbance (General disorders) | 1 | 0 | 2 | 2 | 0 | 0 | 0
Mucosal inflammation (General disorders) | 1 | 0 | 0 | 1 | 0 | 2 | 0
Non-cardiac chest pain (General disorders) | 3 | 1 | 1 | 3 | 0 | 1 | 0
Oedema peripheral (General disorders) | 4 | 3 | 6 | 4 | 5 | 1 | 0
Pyrexia (General disorders) | 5 | 2 | 5 | 5 | 2 | 1 | 2
Bronchitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 2 | 0
Conjunctivitis (Infections and infestations) | 1 | 1 | 3 | 0 | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 1 | 0 | 3 | 0 | 0 | 0
Influenza (Infections and infestations) | 0 | 1 | 1 | 2 | 1 | 1 | 1
Pneumonia (Infections and infestations) | 1 | 1 | 0 | 3 | 0 | 1 | 1
Upper respiratory tract infection (Infections and infestations) | 3 | 2 | 5 | 4 | 3 | 2 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 4 | 0 | 1 | 0 | 2
Fall (Injury, poisoning and procedural complications) | 1 | 4 | 5 | 2 | 1 | 1 | 1
Procedural pain (Injury, poisoning and procedural complications) | 0 | 3 | 2 | 1 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 1 | 2 | 5 | 1 | 2 | 2 | 2
Amylase increased (Investigations) | 2 | 0 | 3 | 1 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 1 | 5 | 2 | 3 | 3 | 2
Blood alkaline phosphatase increased (Investigations) | 1 | 3 | 0 | 0 | 1 | 1 | 1
Blood bilirubin increased (Investigations) | 0 | 0 | 2 | 0 | 2 | 0 | 0
Blood creatinine increased (Investigations) | 5 | 3 | 2 | 0 | 3 | 2 | 2
Lipase increased (Investigations) | 4 | 1 | 3 | 1 | 1 | 0 | 0
Weight decreased (Investigations) | 3 | 1 | 5 | 2 | 1 | 1 | 2
Decreased appetite (Metabolism and nutrition disorders) | 5 | 5 | 12 | 8 | 4 | 5 | 3
Hypercalcaemia (Metabolism and nutrition disorders) | 4 | 2 | 3 | 3 | 1 | 2 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 3 | 1 | 2 | 1 | 3 | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 1 | 3 | 2 | 1 | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 2 | 1 | 1 | 2 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 4 | 0 | 0 | 1 | 1 | 0 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 2 | 1 | 0 | 1 | 1 | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 2 | 1 | 2 | 2 | 0 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 2 | 2 | 1 | 1 | 1 | 2 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 | 1 | 5 | 7 | 7 | 2 | 4
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 5 | 6 | 7 | 6 | 3 | 4
Flank pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 1 | 4 | 2 | 1 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 2 | 2 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0 | 1 | 0 | 2 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 3 | 2 | 6 | 2 | 3 | 2 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 2 | 1 | 5 | 0 | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 2 | 1 | 2 | 1 | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 | 3 | 0 | 5 | 4 | 1 | 2
Amnesia (Nervous system disorders) | 0 | 0 | 2 | 2 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 5 | 3 | 6 | 4 | 2 | 3 | 1
Dizziness postural (Nervous system disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0
Dysgeusia (Nervous system disorders) | 1 | 3 | 1 | 0 | 2 | 1 | 0
Headache (Nervous system disorders) | 4 | 10 | 5 | 1 | 2 | 3 | 3
Lethargy (Nervous system disorders) | 1 | 1 | 1 | 0 | 2 | 0 | 0
Paraesthesia (Nervous system disorders) | 1 | 3 | 1 | 4 | 1 | 2 | 1
Spinal cord compression (Nervous system disorders) | 0 | 2 | 0 | 0 | 1 | 0 | 0
Taste disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 3 | 0 | 0
Tremor (Nervous system disorders) | 2 | 1 | 0 | 1 | 0 | 1 | 0
Anxiety (Psychiatric disorders) | 1 | 3 | 1 | 0 | 1 | 0 | 1
Depression (Psychiatric disorders) | 1 | 2 | 0 | 0 | 2 | 0 | 0
Insomnia (Psychiatric disorders) | 5 | 2 | 4 | 1 | 1 | 2 | 0
Acute kidney injury (Renal and urinary disorders) | 3 | 0 | 0 | 0 | 1 | 1 | 1
Dysuria (Renal and urinary disorders) | 0 | 0 | 3 | 0 | 1 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 2 | 0 | 2 | 1 | 0 | 1 | 0
Urinary retention (Renal and urinary disorders) | 2 | 0 | 0 | 1 | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 11 | 6 | 10 | 8 | 6 | 6 | 2
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 3 | 0 | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 7 | 4 | 6 | 3 | 7 | 2 | 4
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 1 | 0 | 1 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 2 | 0 | 0 | 2 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 1 | 0 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 4 | 1 | 1 | 0 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0 | 0 | 3 | 1 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 1 | 1 | 0 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1 | 0 | 0 | 0 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 4 | 0 | 1 | 1 | 3 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 2 | 1 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 2 | 1 | 2 | 2 | 2 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 2 | 1 | 0 | 1 | 0 | 0 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 3 | 1 | 0 | 3 | 1 | 1 | 1
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 1 | 2 | 1 | 0 | 2 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 10 | 6 | 10 | 8 | 2 | 3 | 1
Rash (Skin and subcutaneous tissue disorders) | 8 | 7 | 12 | 7 | 3 | 4 | 2
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 5 | 1 | 2 | 0 | 0 | 1 | 1
Rash pruritic (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0
Rosacea (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0
Hot flush (Vascular disorders) | 1 | 2 | 1 | 0 | 2 | 0 | 0
Hypertension (Vascular disorders) | 1 | 2 | 4 | 1 | 1 | 2 | 0
Hypotension (Vascular disorders) | 1 | 1 | 2 | 2 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-01-11): https://cdn.clinicaltrials.gov/large-docs/10/NCT02996110/Prot_SAP_000.pdf